CLINICAL TRIAL: NCT02788097
Title: Assessment of Artificial FET Reproductive Outcomes: Transfer of Blastocysts on Progesterone + 4 Versus Progesterone + 5
Brief Title: Comparison of Day 19 and Day 20 Artificial FET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Large and sustained difference in pregnancy rate
Sponsor: Antalya IVF (Other)
Responsible Party: Principal Investigator, Kevin Coetzee, Scientific advisor, Antalya IVF
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AntalyaIVF
Record Dates: First submitted 2016-05-25; First posted 2016-06-02 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Progesterone Induced Endometrial Receptivity
Keywords: blastocysts; progesterone; implantation; artificial frozen embryo transfer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone + 4 (Experimental): the transfer of day 5 blastocyst on the 5th day of progesterone supplementation
  Interventions: Procedure: Progesterone supplementation
- Progesterone + 5 (Active Comparator): the transfer of day 5 blastocysts on the 6th day of progesterone supplementation
  Interventions: Procedure: Progesterone supplementation

INTERVENTIONS:
Procedure: Progesterone supplementation — artificial frozen embryo transfers

SUMMARY:
In recent artificial frozen embryo transfers (FET) in which blastocysts vitrified on day 4 of culture and transferred on P+4, with blastocysts traditionally transferred on P+5, a high rate of implantation has been observed. In addition, a greater number of these implantations resulted in clinical pregnancies (i.e., a conceptus with normal fetal heart activity). In this prospective randomised control study, the investigators will investigate whether this increased viability, is due either to embryo quality, endometrial receptivity, or a combination of the two factors by randomizing the transfer of day 5 blastocysts to P+4 or P+5.

DETAILED DESCRIPTION:
During the first 20 years of IVF embryo transfers were performed on days 1 to 3, even though evidence suggested that embryos dispelled into the uterus from fallopian tubes were at a post-compaction stage. This meant that initially all embryo transfers were asynchronous transfers. This strategy was imposed upon IVF by the vitro culture conditions of the time, which were sub-optimal for normal rates of blastocyst development. Transferred asynchronously cleavage stage embryos have to adapt to "alien" non- physio-metabolic conditions that may result in embryonic stress and compromised embryo development. In fresh embryo transfer this is further exacerbated by the supraphysiological hormone effects of controlled ovarian stimulation. In addition, there are mechanical factors (i.e. uterine contractility) and time factors, related to the endometrium (i.e., window of implantation) and embryo (i.e., time to hatching), that may reduce the chances of implantation. In contrast, to most other mammalian species the transfer of cleavage stage embryos to human uteruses led to acceptable levels of pregnancy and live birth.

The regulation of synchrony between embryo and endometrium has not been fully addressed clinically in the human. This limitation affects IVF significantly in that up to 30% of embryo transfers may be affected by endometrial receptivity factors. The endometrium is a highly specialized, hormonally regulated tissue which is only receptive to embryo communication/interaction for a self-limiting period referred to as the window of implantation. Currently, there is no way to non-invasively determine the time of optimal receptivity, with IVF transfers performed on the assumption that the WOI was sufficiently wide enough to accommodate implantation in most patients and most treatments. During this period, the endometrial epithelium acquires optimal receptivity by progressing through specific structural, functional, and morphological changes induced by pre-ovulatory estrogen and progesterone and post-ovulatory progesterone, LH, and hCG.

During the last three decades, there has been a major increase in the understanding of embryo physiology and correspondingly major improvements in the in vitro culture technologies used, in particular culture media and incubator technologies. These improvements have resulted in the culture of more good quality cleavage stage embryos and consequently blastocysts after extended culture, increasing embryo utility and the pregnancy capacity of an cycle. The increased implantation rates obtained with blastocyst transfers may be as much to do with embryo quality and stage, i.e., blastocysts have the required bi-directional communication competency needed for implantation, as with the WOI, i.e., the time of blastocyst formation and transfer coincides with the WOI of endometria. Moreover, the presently improved culture conditions may also be changing traditional embryo developmental milestones, in particular, the time to blastulation may be decreasing. An increasing number of blastocysts are being formed on day 4 of culture - ±100 hours post-insemination. Traditionally, day 4 embryos were only assessed for evidence of compaction, which is the developmental stage leading to blastulation and cell differentiation.

Zygotes or embryos that reach developmental milestones first (i.e., syngamy, early cleavage, early compaction and early blastulation) are generally believed to have increased chances of normal developmental potential. In recent artificial frozen embryo transfers (FET) in which blastocysts vitrified on day 4 of culture and transferred on P+4, with blastocysts traditionally transferred on P+5, a high rate of implantation has been observed. In addition, a greater number of these implantations resulted in clinical pregnancies (i.e., a conceptus with normal fetal heart activity). In this prospective randomised control study, the investigators will investigate whether this increased viability, is due either to embryo quality, endometrial receptivity, or a combination of the two factors by randomizing the transfer of day 5 blastocysts to P+4 or P+5.

ELIGIBILITY:
Inclusion Criteria:

* a freeze-all cycle

Exclusion Criteria:

* patients who do not consent
* patients who retract their consent
* patients with day 4 blastocysts frozen
* patients with no blastocysts frozen

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya IVF, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
data to be entered

REFERENCES:
- [Background] Fauser BC, Devroey P. Reproductive biology and IVF: ovarian stimulation and luteal phase consequences. Trends Endocrinol Metab. 2003 Jul;14(5):236-42. doi: 10.1016/s1043-2760(03)00075-4. PMID 12826330
- [Background] van de Vijver A, Polyzos NP, Van Landuyt L, Mackens S, Stoop D, Camus M, De Vos M, Tournaye H, Blockeel C. What is the optimal duration of progesterone administration before transferring a vitrified-warmed cleavage stage embryo? A randomized controlled trial. Hum Reprod. 2016 May;31(5):1097-104. doi: 10.1093/humrep/dew045. Epub 2016 Mar 22. PMID 27005893
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone + 4: the transfer of day 5 blastocyst on the 5th day of progesterone supplementation
  Progesterone supplementation: artificial frozen embryo transfers
  61 patients randomized to this group
- Progesterone + 5: the transfer of day 5 blastocysts on the 6th day of progesterone supplementation
  Progesterone supplementation: artificial frozen embryo transfers
  69 patients randomized to this group
Period: Overall Study
Arm/Group | Progesterone + 4 | Progesterone + 5
Started | 61 | 69
Completed | 61 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone + 4 | Progesterone + 5 | Total
Number analyzed (Participants) | 61 | 69 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 69 | 130
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (4.3) | 28.5 (3.2) | 28.35 (3.75)
Gender [Count of Participants; unit: Participants]
  Female | 61 | 69 | 130
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 61 | 69 | 130

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Pregnancy
Description: >30IU/L of serum βhCG on day 14 of cycle
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Progesterone + 4 | Progesterone + 5
Number analyzed (Participants) | 61 | 69
percentage of participants | 52.5 | 79.7

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Progesterone + 4 | Progesterone + 5
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/69
Other Adverse Events (participants affected / at risk) | 0/61 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes